CLINICAL TRIAL: NCT04036799
Title: Development of a Risk Calculator to Predict Sudden Cardiac Death in Children With Hypertrophic Cardiomyopathy
Brief Title: PRecIsion Medicine in CardiomyopathY
Acronym: PRIMaCY
Status: Active, not recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Stanford University (Other); Children's Hospital of Philadelphia (Other); New York Presbyterian Hospital (Other); University of Texas Southwestern Medical Center (Other); University of Michigan (Other); Children's Hospital Medical Center, Cincinnati (Other); Provincial Health Services Authority British Columbia (Other); Stollery Children's Hospital (Other); Children's Hospital of Eastern Ontario (Other); Royal Children's Hospital (Other); Children's Healthcare of Atlanta (Other); Primary Children's Hospital (Other); Baylor College of Medicine (Other); The Cleveland Clinic (Other); Monroe Carell Jr. Children's Hospital at Vanderbilt (Other); Children's Hospital Colorado (Other); Indiana University Health (Other); OHSU Doernbecher Children's Hospital (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Seema Mital, Principal Investigator, The Hospital for Sick Children
Other Study IDs: 1000055819
Record Dates: First submitted 2019-07-23; First posted 2019-07-30 (Actual); Results first posted 2021-03-11 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Hypertrophic Cardiomyopathy; Sudden Cardiac Death
Keywords: Pediatric; Risk Prediction
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertrophic Cardiomyopathy

SUMMARY:
This is a retrospective cohort study of pediatric hypertrophic cardiomyopathy (HCM) patients using chart and registry review methodology. The studies objective is to develop and validate a sudden cardiac death (SCD) risk calculator that is age-appropriate for children with HCM that includes clinical and genetic factors.

ELIGIBILITY:
Inclusion Criteria:

* phenotype-positive patients diagnosed with hypertrophic cardiomyopathy
* phenotype-negative, genotype positive patients considered at risk for developing hypertrophic cardiomyopathy

Exclusion Criteria:

* Neuromuscular, metabolic, syndromic (other than Noonan Syndrome and related RAS-opathies) or endocrine (including infants of diabetic mothers) causes of HCM
* (Other treatable causes of left ventricular hypertrophy (systemic hypertension, anatomic defects causing left ventricular outflow tract obstruction e.g. aortic stenosis, subAS, subaortic membrane, coarctation)

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals meeting eligibility criteria at first presentation were included.
Sampling Method: Non-Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2026-12 (Estimated)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Miron A, Lafreniere-Roula M, Steve Fan CP, Armstrong KR, Dragulescu A, Papaz T, Manlhiot C, Kaufman B, Butts RJ, Gardin L, Stephenson EA, Howard TS, Aziz PF, Balaji S, Ladouceur VB, Benson LN, Colan SD, Godown J, Henderson HT, Ingles J, Jeewa A, Jefferies JL, Lal AK, Mathew J, Jean-St-Michel E, Michels M, Nakano SJ, Olivotto I, Parent JJ, Pereira AC, Semsarian C, Whitehill RD, Wittekind SG, Russell MW, Conway J, Richmond ME, Villa C, Weintraub RG, Rossano JW, Kantor PF, Ho CY, Mital S. A Validated Model for Sudden Cardiac Death Risk Prediction in Pediatric Hypertrophic Cardiomyopathy. Circulation. 2020 Jul 21;142(3):217-229. doi: 10.1161/CIRCULATIONAHA.120.047235. Epub 2020 May 18. PMID 32418493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter retrospective observational cohort study of pediatric patients with clinically diagnosed childhood-onset HCM. The primary cohort included patients from 11 sites participating in the PRIMaCY study (Precision Medicine for Cardiomyopathy), an international registry of patients with pediatric HCM launched in 2017. These included 4 Canadian, 6 US, and 1 Australian site. For model validation, we used data from the Sarcomeric Human Cardiomyopathy Registry.
Groups:
- Hypertrophic Cardiomyopathy: Patients with a clinical diagnosis of HCM defined as having an LV posterior wall or septal thickness z score ≥2.
Period: Overall Study
Arm/Group | Hypertrophic Cardiomyopathy
Started | 572
Completed | 572
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants with a clinical diagnosis of HCM
Groups:
- Hypertrophic Cardiomyopathy: Patients included were those with a clinical diagnosis of HCM defined as having LV posterior wall or septal thickness z score ≥2, age <18 years at the time of diagnosis, absence of a SCD event before diagnosis, and at least 1 follow-up assessment after diagnosis.
Arm/Group | Hypertrophic Cardiomyopathy
Number analyzed (Participants) | 572
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 9.8 [2.1 to 13.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178
  Male | 394
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 235
  Canada | 273
  Australia | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Composite Sudden Cardiac Death Event
Description: The composite SCD event includes post diagnosis SCD, aborted SCD (including ventricular fibrillation, sustained ventricular tachycardia), primary ICD insertion with appropriate shock, secondary ICD insertion
Time Frame: Time to a composite sudden cardiac death event during 5-year follow-up
Population: Patients with a clinical diagnosis of HCM defined as having an LV posterior wall or septal thickness z score ≥2, age <18 years at the time of diagnosis, absence of a sudden cardiac death event before diagnosis, and at least 1 follow-up assessment after diagnosis.
Measure: Count of Participants; unit: Participants
Groups:
- Hypertrophic Cardiomyopathy: Phenotype-positive HCM diagnosed between 1987 and 2018
Arm/Group | Hypertrophic Cardiomyopathy
Number analyzed (Participants) | 572
Participants | 53
Statistical Analysis 1: Comparison: Hypertrophic Cardiomyopathy; Test type: Other — Categorical variables were summarized using frequencies and proportions; Cumulative proportion of events at 5 yrs = 9.1

ADVERSE EVENTS:
Description: Adverse events were not captured as this was a retrospective observational cohort study
Arm/Group | Hypertrophic Cardiomyopathy
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study has limitations inherent to any retrospective analysis, that includes missing data, survivor bias, and lower uptake of genetic testing in the earlier era. Missing echocardiographic data were addressed through a re-review of echocardiograms where available and through imputation where this was not possible. We deliberately did not perform an echocardiographic core laboratory analysis because a real-world, point-of-care tool has to rely on locally acquired data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT04036799/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT04036799/SAP_001.pdf